CLINICAL TRIAL: NCT05377619
Title: Gastric Glitch: a New Functional Disease Treated With Prucalopride and Buspirone in a N-of-1 Double-blind Clinical Trial
Brief Title: Preventing Gastric Glitch With Prucalopride and Buspirone: N-of-1 Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Responsible Party: Principal Investigator, Fernando Fornari, Professor, Universidade de Passo Fundo
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 5.151.164
Record Dates: First submitted 2022-04-20; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — prucalopride; Buspirone

STUDY DESIGN:
Intervention Model Description: N-of-1 trial testing the effect of prucalopride, buspirone and placebo on the prevention of alcohol-induced gastric glitch
Who Masked: Participant, Investigator
Masking Description: Identical capsules containing prucalopride, buspirone or placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- prucalopride (Experimental): prucalopride 2 mg 1 capsule orally 1 hour before the wine challenging (during a dinner), in five dinners (2 dinners per week)
  Interventions: Drug: Prucalopride
- buspirone (Experimental): buspirone 10 mg 1 capsule orally 1 hour before the wine challenging (during a dinner), in five dinners (2 dinners per week)
  Interventions: Drug: Buspirone
- placebo (Placebo Comparator): placebo 1 capsule orally 1 hour before the wine challenging (during a dinner), in five dinners (2 dinners per week)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — prucalopride 2 mg 1 hour before the challenge with intake of wine (200 ml) and a dinner
  Other Names: Resolor
  Arms: prucalopride
Drug: Buspirone — buspirone 10 mg 1 hour before the challenge with intake of wine (200 ml) and a dinner
  Other Names: Ansitec
  Arms: buspirone
Drug: Placebo — placebo 1 hour before the challenge with intake of wine (200 ml) and a dinner
  Arms: placebo

SUMMARY:
Background: Gastric glitch is a new functional disease characterized by severe and transient epigastric pain occurring after challenges such as drinking alcohol and eating specific foods. Aims: In this N-of-1 trial, we first characterized the clinical and gastric tomographic images of a patient with gastric glitch highly reproducible after alcohol challenging, and then tested the effect of prucalopride and buspirone on the prevention of gastric glitch crises.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of prucalopride and buspirone, compared to placebo, in the prevention of gastric pain crises, in a double-blind clinical trial of a single patient. Methods: Female, 35 years old, with signed consent to participate in the study, received 15 capsules to take 1 capsule 60 minutes before ingesting 200 ml of red wine at home (≈20 grams of alcohol), twice a week, according to her routine food, totaling 15 meals. Thus, the experimental phase lasted about eight weeks. The 15 capsules contain placebo (5 capsules), prucalopride 2 mg (5 capsules) or buspirone 10 mg (5 capsules), prepared by a specialized pharmacy in such a way that their physical characteristics do not allow the identification of which agent is being administered, neither by the patient nor the investigator controlling the trial (double-blind). The aforementioned pharmacy generated a code for each pill, randomly, and provided a sealed list with the 15 codes and their respective drugs, for disclosure after the end of the study. The patient was instructed to record in a standardized diary the occurrence of pain crises after the wine challenge, as well as their duration and intensity (Likert 0 to 10: maximum pain), and accompanying symptoms. The patient was asked to contact the researchers directly (WhatsApp) throughout the trial, to clarify any doubts or need for some assistance due to the occurrence of symptoms related to the study. The study statistics will be descriptive in terms of pain events, and the effect of the drugs will be evaluated in a statistical model suitable for the N-of-1 trial. Prucalopride is a 5-HT4 receptor agonist that accelerates gastric emptying, while buspirone is a 5-HT1A receptor agonist that enhances gastric accommodation function. The presumed pathophysiology underlying the patient's pain is retention of wine in the gastric lumen, causing pain. Stimulating gastric emptying with prucalopride or increasing the accommodation of the gastric fundus with buspirone could prevent or alleviate the pain crisis.

ELIGIBILITY:
Inclusion Criteria:

* adult patient suffering from severe gastric pain after ingestion of a small amount of wine

Exclusion Criteria:

* N/A (N-of-1 trial)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Pain severity during gastric glitch crises | 2 hours after challenging with wine intake
  Pain severity scored by the patient using a Likert scale (1 = minimal / 10 = maximal pain) following wine intake (200 ml)

OTHER OUTCOMES:
Occurrence of side effects secondary to tested drugs | 12 hours after drugs intake
  Registration by the patient (symptom diary) concerning the occurrence (yes/not) of side effects potentially related with prucalopride (abdominal cramps, nausea, diarrhea, and headache) and buspirone (drowsiness and dizziness) after each ethylic challange

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fornari, Principal Investigator — University of Passo Fundo
Locations (1):
- University of Passo Fundo, Passo Fundo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No